CLINICAL TRIAL: NCT00430924
Title: The Effect of Aldosterone Inhibition on Proteinuria in Patients With Progressive Renal Disease
Brief Title: Inhibition of Aldosterone in Patients With Chronic Renal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lene Boesby (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Lene Boesby, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B109LB1; 2006-004411-21
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney Failure, Chronic; Proteinuria; Aldosterone; Renin-Angiotensin System
MeSH Terms: conditions — Kidney Failure, Chronic; Proteinuria | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Eplerenone
  Interventions: Drug: Eplerenone
- 2 (No Intervention): Control
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Once daily administration for 8 weeks and 8 weeks control.

SUMMARY:
The purpose of this study is to examine whether the inhibition of aldosterone will result in lower excretion of protein via urine. The hypothesis is that if loss of protein is lowered, progression of renal disease with be slower than otherwise expected.

DETAILED DESCRIPTION:
Patients with chronic renal disease are likely to progress to end stage renal disease with the need for renal replacement therapy. It is accepted that proteinuria is a surrogate measurement for progression. If proteinuria can be lowered we hope to prolong patients pre-dialysis phase. Our theory is that aldosterone inhibition will lead to this.

For a period of 8 weeks patients will be randomized to either aldosterone receptor inhibition with the drug eplerenone or control without. Blood pressures will be kept at the same level using other drugs.

ELIGIBILITY:
Inclusion Criteria:

* Proteinuria > 500 mg/24 hours
* Hypertension or anti-hypertensive treatment

Exclusion Criteria:

* Diabetic nephropathy
* GFR< 20 ml/min
* P-potassium between 3,5 mmol/l and 5,0 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Proteinuria reduction | bi-monthly

SECONDARY OUTCOMES:
Evaluating blood pressure response and hyperkalaemia after aldosterone inhibition. | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Svend Strandgaard, DMSc, Study Director; Anne-Lise Kamper, DMSc, Study Director — nonaffiliated
Locations (2):
- Denmark (2):
  - Rigshospitalet, Blegdamsvej 9, Copenhagen
  - Herlev Hospital, Herlev

REFERENCES:
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Boesby L, Elung-Jensen T, Klausen TW, Strandgaard S, Kamper AL. Moderate antiproteinuric effect of add-on aldosterone blockade with eplerenone in non-diabetic chronic kidney disease. A randomized cross-over study. PLoS One. 2011;6(11):e26904. doi: 10.1371/journal.pone.0026904. Epub 2011 Nov 4. PMID 22073219
- See also: Publication — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0026904